CLINICAL TRIAL: NCT00641576
Title: A Study to Evaluate the Morse Taper Lock and Connection of the ACE Implant Internal-Connection and Its Effect of the Biological Gap
Brief Title: Evaluation of the ACE Dental Implant
Acronym: ACE-2005
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: ACE Surgical Supply, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Reddy, DMD, Interin Dean, University of Alabama at Birmingham
Other Study IDs: W050404001
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Edentulism
Keywords: Endosseous implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ACE CONNECT Endosseous dental implant — Subjects in this study receive ACE CONNECT Internal-Connection dental implants to: 1)replace a missing tooth in an edentulous area of the maxilla or mandible restored with a single-unit crown (may include up to two non-adjacent areas as study sites) or, 2)subjects with an edentulous mandible will receive two implants placed in the lower canine position and restored with an implant-retained removable over-denture.
  Subjects will return for four follow-up evaluations scheduled at 6, 12, 18 and 24 months after delivery of the permanent restoration.
  Other Names: ACE Morse Taper Lock; ACE Implant Internal-Connection

SUMMARY:
Dental implants are small metal posts that look like miniature screws. They are surgically implanted into the jawbone where they serve as substitute tooth roots. Implants are used in dentistry to reestablish function and aesthetics to areas of the mouth were natural teeth are missing.

Classical dental implants are made in two pieces. One part anchors in the jawbone and one part serves as a connecting post (an abutment) that attaches to a crown restoration or to attachment clasps that hold a denture in place.

Occasionally the materials used to fasten the two implant components together work their way loose and over time the abutment may begin to disconnect. If this happens a small gap appears between the implant and abutment. There are many reasons why this loosening occurs. One reason may be the design of the implant itself and another may be the way the two components are fastened together.

This study will assess the performance of an implant with a new design. The investigators hypothesize that using this implant design will reduce the risk of an implant-abutment disconnect and improve long-term success of implant therapy.

DETAILED DESCRIPTION:
While the external hex dental implant design has had very good clinical success, it is limited by retention screw loosening at the junction of the implant fixture and abutment; a situation that leads to micro-movement between components.

A number of clinical complications may arise when implant components separate. Micro-movement between the implant abutment and seating platform is thought to contribute to the formation of a "biological gap", the most notable consequence being gradual resorption of crestal alveolar bone over time.

We hypothesize that the "ACE CONNECT" two-piece implant design with an internal connection will limit screw loosening by providing a stable junction between the body of the implant and the abutment; a more stable junction will limit micro-movement and prevent the formation of a gap between components. Limiting the gap will lead to less inflammation of peri-implant soft tissues and reduced resorption of bone adjacent to the implant.

ELIGIBILITY:
Inclusion Criteria:

* Need for replacement of non-adjacent missing teeth with dental implants
* Edentulous in the area for more than 2 months
* Minimum native bone height and width to receive a 10mm X 4mm implant

Exclusion Criteria:

* Untreated decay or periodontal disease in residual dentition
* Need for bone or soft-tissue augmentation in the proposed implant site
* Pregnancy
* Consistent use of medications likely to compromise bone healing
* Chronic disease condition likely to compromise bone healing
* Consistent smoking over 10 cigarettes during the immediate past 6 months

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental school periodontology clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2005-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Junctional stability between device and abutment | 24 months

SECONDARY OUTCOMES:
Peri-implant osseous support of the device | 24 months
Peri-implant soft-tissue response to the device | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Reddy, DMD, DMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama, United States

REFERENCES:
- [Background] Zarb GA, Schmitt A. The longitudinal clinical effectiveness of osseointegrated dental implants: the Toronto study. Part III: Problems and complications encountered. J Prosthet Dent. 1990 Aug;64(2):185-94. doi: 10.1016/0022-3913(90)90177-e. PMID 2202818
- [Background] Goodacre CJ, Kan JY, Rungcharassaeng K. Clinical complications of osseointegrated implants. J Prosthet Dent. 1999 May;81(5):537-52. doi: 10.1016/s0022-3913(99)70208-8. PMID 10220658
- [Background] Jemt T, Book K, Linden B, Urde G. Failures and complications in 92 consecutively inserted overdentures supported by Branemark implants in severely resorbed edentulous maxillae: a study from prosthetic treatment to first annual check-up. Int J Oral Maxillofac Implants. 1992 Summer;7(2):162-7. PMID 1398832
- [Background] Naert I, Quirynen M, van Steenberghe D, Darius P. A study of 589 consecutive implants supporting complete fixed prostheses. Part II: Prosthetic aspects. J Prosthet Dent. 1992 Dec;68(6):949-56. doi: 10.1016/0022-3913(92)90557-q. PMID 1494126
- [Background] Kallus T, Bessing C. Loose gold screws frequently occur in full-arch fixed prostheses supported by osseointegrated implants after 5 years. Int J Oral Maxillofac Implants. 1994 Mar-Apr;9(2):169-78. PMID 8206552
- [Background] Jemt T, Laney WR, Harris D, Henry PJ, Krogh PH Jr, Polizzi G, Zarb GA, Herrmann I. Osseointegrated implants for single tooth replacement: a 1-year report from a multicenter prospective study. Int J Oral Maxillofac Implants. 1991 Spring;6(1):29-36. PMID 1843491
- [Background] Becker W, Becker BE. Replacement of maxillary and mandibular molars with single endosseous implant restorations: a retrospective study. J Prosthet Dent. 1995 Jul;74(1):51-5. doi: 10.1016/s0022-3913(05)80229-x. PMID 7674191
- [Background] Lazzara R, Siddiqui AA, Binon P, Feldman SA, Weiner R, Phillips R, Gonshor A. Retrospective multicenter analysis of 3i endosseous dental implants placed over a five-year period. Clin Oral Implants Res. 1996 Mar;7(1):73-83. doi: 10.1034/j.1600-0501.1996.070109.x. PMID 9002825
- [Background] Binon PP. Evaluation of the effectiveness of a technique to prevent screw loosening. J Prosthet Dent. 1998 Apr;79(4):430-2. doi: 10.1016/s0022-3913(98)70157-x. PMID 9576318
- [Background] McGlumphy EA, Mendel DA, Holloway JA. Implant screw mechanics. Dent Clin North Am. 1998 Jan;42(1):71-89. PMID 9421671
- [Background] Hurson S. Laboratory techniques to prevent screw loosening on dental implants. J Dent Technol. 1996 Apr;13(3):30-7. PMID 9516271
- [Background] Bragger U, Hafeli U, Huber B, Hammerle CH, Lang NP. Evaluation of postsurgical crestal bone levels adjacent to non-submerged dental implants. Clin Oral Implants Res. 1998 Aug;9(4):218-24. doi: 10.1034/j.1600-0501.1998.090402.x. PMID 9760896
- [Background] Weber HP, Buser D, Fiorellini JP, Williams RC. Radiographic evaluation of crestal bone levels adjacent to nonsubmerged titanium implants. Clin Oral Implants Res. 1992 Dec;3(4):181-8. doi: 10.1034/j.1600-0501.1992.030405.x. PMID 1298433
- [Background] Lekholm U, Zarb G. Patient selection and preparation. In Branemark P-I, Zarb GA and Albrektsson T. eds. Tissue Integrated Prosthesis: Osseointegration in Clincal Dentistry. Chicago: Quintessence 1985 pp 199-209